CLINICAL TRIAL: NCT04206267
Title: The Effectiveness of Vibrational Applications On Orthodontic Treatment: A Randomized-Controlled Clinical Trial
Brief Title: The Effectiveness of Vibrational Applications on Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Baris Can Telatar, Principal investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 709045004/134
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Control Group; Acceledent Group
Keywords: Tooth movement; AcceleDent; distalizing

STUDY DESIGN:
Intervention Model Description: Subjects were randomly allocated to either the AcceleDent group or the control group. The randomization was achieved by coin-tossing by one investigator. This method is equivalent to tossing a coin for each subject that enters a trial, such as Heads = control group, Tails = AcceleDent group.
Who Masked: Investigator
Masking Description: One investigator assigned the patients to study or control group and conducted the linear measurements with 3D Trios System, other investigator treated the samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceledent group (Experimental): Patients up to 18 years old who were planned first premolar extractions assigned to study group. AcceleDent Aura appliance was applied for 20 minutes per day. during canine retraction.
  Interventions: Device: Acceledent
- Control group (No Intervention): Patients up to 18 years old who were planned first premolar extractions assigned to control group. The canine retractions were performed without any additional vibrational device.

INTERVENTIONS:
Device: Acceledent — Device for accelerating tooth movement
  Arms: Acceledent group

SUMMARY:
The aim of this study is to determine whether vibrational applications, as an adjunct to orthodontic forces, increases the rate of tooth movement in patients with fixed orthodontic appliances.

DETAILED DESCRIPTION:
Nineteen patients who had class 2 division 1 malocclusion or severe crowding and needed first premolar extractions as a treatment modality were included to the study. The patients were divided into two groups, 8 in control and 11 in the study. The subjects assigned to study group were applied suplementary vibrational forces for 20 min/daily. 3-dimensional digital models were generated just before canine distalization and after space closure by 3Shape TRİOS R700 (3Shape Inc., Copenhagen, Denmark) device. The linear measurements between molars and canines were evaluated. The results were assessed with SPSS 23.0 programme (lBM SPSS Statistics for Windows, NY, USA). The amount of tooth movement for all samples were measured twice by the responsible investigator at one week interval. Interclass correlation coefficient-ICC was used to asses intraobserver accuracy and reliability.Mann- Whitney U test was used to assess treatment effect in terms of time to reach canine distalization. Correlation between measurements were described with Spearman Correlation Coefficient. Interclass correlation was 95%, which is in the range of excellent measurement agreement.

ELIGIBILITY:
Inclusion Criteria:

* patients who were planned first premolar extractions
* demonstrated good oral hygiene

Exclusion Criteria:

* patients with poor oral hygiene and have periodontal problem

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
canine retraction rate | 6 months
  İnitial measurements were conducted after levelling stage and prior to retraction of the canine tooth. Linear measurements were performed between mesial edges of molar tubes and distal edges of canine brackets. Due to using TADs as direct anchorage it is considered that the molars remained constant during the retraction process. After retraction stage, measurements were performed between the mesial edges of the molar tubes and the distal edges of the canine brackets, and the monthly tooth movement rates were detected according to the difference between initial and second measurements.

SECONDARY OUTCOMES:
the compliance data on device use | 6 months
  it was collected by downloading the tracking information on the device

CONTACTS AND LOCATIONS:
Overall Officials: Baris Telatar, Principal Investigator — Akdeniz University Department of Orthodontics

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study submission to journal

REFERENCES:
- [Background] Woodhouse NR, DiBiase AT, Johnson N, Slipper C, Grant J, Alsaleh M, Donaldson AN, Cobourne MT. Supplemental vibrational force during orthodontic alignment: a randomized trial. J Dent Res. 2015 May;94(5):682-9. doi: 10.1177/0022034515576195. Epub 2015 Mar 10. PMID 25758457